CLINICAL TRIAL: NCT06169241
Title: Effect of Nitrate Supplementation on Blood Pressure and Systemic Microvascular Function of Resistant Hypertensive Patients
Brief Title: Effect of Nitrate Supplementation on Blood Pressure and Microvascular Function of Resistant Hypertensive Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Cardiology, Laranjeiras, Brazil (Other Government)
Responsible Party: Principal Investigator, Eduardo Tibirica, MD, PhD, Senior Researcher, National Institute of Cardiology, Laranjeiras, Brazil
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 70847523.9.0000.5272
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Arterial Hypertension; Resistant Hypertension; Microvascular Function; Nitrate Supplementation
Keywords: microcirculation; capillary density; microvascular reactivity; systemic resistant hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Treatment with beetroot extract powder - nutritional supplementation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): The placebo group will be administered as a colored and flavored isocaloric supplement composed of maltodextrin.
  Interventions: Dietary Supplement: Placebo
- Beetroot extract (Active Comparator): Beetroot extract powder supplementation with 400mg of nitrate per dose in the amount of 10g per day orally will be used in the group.
  Interventions: Dietary Supplement: Beetroot extract

INTERVENTIONS:
Dietary Supplement: Beetroot extract — Beetroot extract powder supplementation with 400mg of nitrate per dose in the amount of 10g per day orally will be used in the group.
  Arms: Beetroot extract
Dietary Supplement: Placebo — The placebo will be administered as a colored and flavored isocaloric supplement composed of maltodextrin.
  Arms: Placebo

SUMMARY:
Arterial hypertension (AH) has been identified as an important public health problem and considered a new epidemic with high mortality and morbidity. High blood pressure (BP) levels increase the chances of coronary artery disease (CAD), heart failure (HF), stroke, chronic renal failure (CRF) and death. Beetroot powder may be an easier way to increase the availability of nitric oxide and consequently vasodilation in these patients. However, studies are needed to evaluate its benefits in patients with AH.

ELIGIBILITY:
Inclusion Criteria:

* Resistant hypertension, with a diagnosis described in the medical record, without changing medications or increasing doses in the last 30 days.

Exclusion Criteria:

* neoplasms
* heart failure
* use of medications with nitrate in their formula
* patients undergoing renal denervation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of blood pressure evolution | 60 days
  Evaluation using Ambulatory Blood Pressure Monitoring: systolic, diastolic and mean arterial pressures

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Cardiology, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No